CLINICAL TRIAL: NCT00859365
Title: Efficacy of an Integrative Approach Utilizing Acupuncture as an add-on Therapy for the Treatment of Back and Neck Pain in an Emergency Department Setting - A Comparative Randomized Controlled Trial
Brief Title: Acupuncture for Back and Neck Pain in an Emergency Room Setting
Acronym: ABNP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Head of Emergency Department, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 127/08
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Back Pain; Neck Pain; Anxiety; Range of Motion
Keywords: back pain; neck pain; anxiety; range of motion
MeSH Terms: conditions — Back Pain; Neck Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acupuncture (Experimental): Real Acupuncture
  Interventions: Procedure: Real Acupuncture
- 2 Placebo acupuncture (Placebo Comparator)
  Interventions: Procedure: Placebo Acupuncture
- 3 No treatment (No Intervention): No treatment performed
  Interventions: Procedure: No intervention

INTERVENTIONS:
Procedure: Real Acupuncture — Real acupuncture treatment in real acupuncture points
  Arms: Acupuncture
Procedure: Placebo Acupuncture — empty plastic acupuncture guide-tube located on the patients back in a non visable area and connected to a visible electric stimulator
  Arms: 2 Placebo acupuncture
Procedure: No intervention — Patients lay down for a period of 35 minutes without any treatment o intervention
  Arms: 3 No treatment

SUMMARY:
This study aims to examine the efficacy of an Integrative approach utilizing Acupuncture as an add-on therapy for the treatment back and neck pain in an emergency department setting

Acupuncture is well established as an effective treatment for back pain. The investigators cumulative experience in Asaf Harofeh Medical Center has shown Acupuncture to be an Effective therapy for simple back and neck pain in an ER setting.

This study will examine weather Acupuncture can decrease pain, increase range of motion and decrease anxiety in patients admitted to the Emergency Room with simple back and neck pain without neurological findings. Acupuncture will be performed as an add on therapy on top of analgesic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and females age 18-60 with acute or sub acute/chronic simple back or neck pain
* Agreed to a physical examination and by an orthopedic physician and X-ray
* Diagnosis of simple back pain with levels of 4<NRS at least
* Agreed and able to fill pain, anxiety and satisfactory questioners
* Agreed and able to sign informed consent

Exclusion Criteria:

* Fracture, sprain or neurological deficit during physical examination
* Pain scale of NRS< 4
* Referred or radiating pain
* Active pregnancy
* Active inflammatory arthritis
* History of CVA
* Open wounds
* Acute malignancy with life expectancy of less than 5 years
* Experience with acupuncture treatments
* History of drug addiction
* History of osteoporosis
* Declined or unable to sign informed consent
* Soldiers in active military service

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2009-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
A comparable difference in pain levels between a combined medication and acupuncture treatment to medication treatment alone as measured by the Numeric Rating Scale (NRS) | At day of treatment, after 24 hrs

SECONDARY OUTCOMES:
4.2.1 A comparable difference in range of motion between a combined medication and acupuncture treatment to medication treatment alone as measured by Spine Scan Device and physical exam using gonoimeter | day of treatment, after 24 hrs
4.2.2 A comparable difference in patient self reported anxiety assessed by Hebrew version of the anxiety and somatization sections of the Symptom Check List-90 questioner (SCL-90) | day of treatment
4.2.3 A comparable difference in the amount of analgesic pain medication consumed by the patients during the week following the treatment | day of treatment and after 24 hours
4.2.4 A comparable difference in safety and patient satisfactory as measured by overall satisfactory and safety questionnaires | day of treatment, after 1 weekl

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Bar-Haim, MD, Principal Investigator — Asaf Harofeh Medical Center, Zerifin, Israel; Amos Ziv, M.Sc, Study Director — Asaf Harofeh Medical Center
Locations (1):
- Asaf Harofeh Medical Center, Beer-Yaacob, Zerifin, Israel, Israel